CLINICAL TRIAL: NCT04128605
Title: Suprascapular Nerve Block Versus Intraarticular Steroid Injection in Hemiplegic Shoulder Pain: A Randomized Double Blinded Control Trial
Brief Title: Suprascapular Nerve Block Versus Intraarticular Steroid Injection in Hemiplegic Shoulder Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Anwar Suhaimi, Senior Lecturer and Rehabilitation Physician, University of Malaya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201945-7301
Record Dates: First submitted 2019-09-10; First posted 2019-10-16 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Hemiplegic Shoulder Pain

STUDY DESIGN:
Intervention Model Description: 1. Patients referred to Rehabilitation Clinic for hemiplegic shoulder pain (HSP) will be recruited.
  2. Patients will be randomly allocated using a computer program into suprascapular nerve block (SSNB) (Intervention) vs intra-articular shoulder steroid injection (IAS) (Control) group
  3. Intervention Group
     SSNB performed by skilled interventionist who is not blinded for safety reason 5 mls of Bupivacaine, 5 mls Lidocaine and 10 mls of saline
  4. Control group
     IAS performed by skilled interventionist who is blinded on patient's initial measurement 40 mg of Triamcinolone Acetate + 2 ml of Lidocaine 1%
  5. Evaluations will be repeated at:
     * 1 hour, 1 month and 3 months for maximum (max) passive range of motion (PROM), numerical rating scale (NRS) at max PROM
     * 1 month and 3 months for shoulder disability questionnaire (SDQ) and shoulder pain and disability index (SPADI)
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded from knowing the intervention they're receiving.
  Both suprascapular nerve block and intraarticular shoulder steroid injection will be performed at posterior aspect of shoulder while participant is in seated position and facing forward.
  The assessor will also be blinded from knowing which group the participants belong to.
  All the medical record related to this study will be inaccessible by the assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention: Suprascapular nerve block (SSNB) (Experimental): SSNB performed by skilled interventionist who is not blinded for safety reason. 5 mls of Bupivacaine, 5 mls Lidocaine and 10 mls of saline.
  Interventions: Procedure: Suprascapular nerve block (SSNB)
- Control: Intraarticular shoulder steroid injection (IAS) (Active Comparator): IAS performed by skilled interventionist who is blinded on patient's initial measurement.
  40 mg of Triamcenolone Acetate + 2 ml of Lidocaine 1%
  Interventions: Procedure: Intraarticular shoulder steroid injection (IAS)

INTERVENTIONS:
Procedure: Suprascapular nerve block (SSNB) — SSNB is performed using ultrasound guidance by skilled interventionist under ultrasound guidance.
  Skin area at posterior shoulder is first infiltrated with Lidocaine 1%. Then, a mixture of 5 mls of Bupivacaine, 5 mls Lidocaine 1% and 10 mls of saline are injected at posterior shoulder towards suprascapular notch surrounding suprascapular nerve.
  Arms: Intervention: Suprascapular nerve block (SSNB)
Procedure: Intraarticular shoulder steroid injection (IAS) — IAS is performed using ultrasound guidance by skilled interventionist under ultrasound guidance.
  Skin area at posterior shoulder is first infiltrated with Lidocaine 1%. IAS is performed by injecting 40 mg of Triamcenolone Acetonide along with 2 ml of Lidocaine 1% into glenohumeral articular space
  Arms: Control: Intraarticular shoulder steroid injection (IAS)

SUMMARY:
Suprascapular nerve block versus(vs) intra-articular steroid injection in the management of hemiplegic shoulder pain (HSP): a randomised, double blinded, controlled trial

BACKGROUND Hemiplegic shoulder pain (HSP) is a common complication of stroke. It can happen as early as one week post stroke with a frequency as high as 72%. HSP can result in significant disability as pain and limited shoulder range of motion (ROM) decrease hand function, reduce participation in rehabilitation activity and delay functional recovery of the patients. Management of HSP focused on reducing pain and improving shoulder ROM. Minimally invasive treatment of HSP with intra-articular shoulder steroid (IAS) injection and supra-scapular nerve block (SSNB) have gained interest.

OBJECTIVES

Primary objective:

1. To assess the analgesic effect of SSNB vs IAS in HSP among Malaysian stroke population.

   Secondary objectives:
2. To assess the improvement of passive ROM post SSNB versus IAS in HSP.
3. To assess for improvement of functional outcome post SSNB versus IAS in HSP.

METHOD

A prospective, double blinded interventional study will be conducted in the Rehabilitation Medicine Clinic, University of Malaya Medical Centre for a duration of 1 year. Eligible subjects will be enrolled from all referrals of hemiplegic shoulder pain (HSP), following computer-generated randomization they will be allocated to either supra-scapular nerve block (SSNB) (intervention) or intra-articular shoulder steroid injection (IAS) (control) groups. The subjects and assessors are blinded to the intervention received, which will be performed by an experienced interventionist, not participating in randomization or data collection and analysis. Demographics of participants time since stroke, etiology, presence of spasticity, Numerical Rating Score (NRS) pain score at maximal passive ROM, maximum passive ROM of shoulder flexion, abduction, internal and external rotation as well as SDQ and SPADI will recorded prior to injection, 1 hour, 1 month and 3 months post injection. Mann-Whitney U tests and Chi-Square test of association will be used as appropriate to compare groups at baseline. Shoulder ROM and NRS pre and post intervention will be analysed using paired t-test and ANOVA. Functional outcome of SDQ and SPADI pre and post intervention will be analysed using paired t-test as well.

DETAILED DESCRIPTION:
1. INTRODUCTION

1.1 Research Area

Hemiplegic shoulder pain (HSP) is a common clinical consequence of stroke with reported frequency as high as 72% (1). Onset of HSP is more common at 2-3 months post stroke(2). HSP can reduce participation in rehabilitation activities and reduce quality of life(3). The etiology of HSP includes neurological and mechanical factors, although mechanical factors are more common. Mechanical factors include structural injury from glenohumeral subluxation, or rotator cuff pathology (3). In hemiplegic patients, the nociceptive pain ratio was higher at 86.7% compared to neuropathic pain ratio; 13.3% (4). Management of HSP focused on reducing pain and improving shoulder ROM. Minimally invasive treatment of HSP with intra-articular steroid (IAS) injection and supra-scapular nerve block (SSNB) have lately gained interest. However, 2 studies done so far showed that while both SSNB and IAS showed significant differences in reducing shoulder pain and improving ROM with time, there was no significant difference of these injection method in comparison to conventional treatment. None of the studies done to date documents functional outcome of patients post injection with IAS or SSNB. The main purpose of this study is to assess the analgesic effect of SSNB vs IAS in HSP among Malaysian stroke population as well as to look at the improvement of shoulder ROM and functional outcome measure.

1.2 Research Questions

Does supra-scapular nerve block (SSNB) provide better pain relief, passive range of motion (PROM) and functional outcome compared to intraarticular steroid (IAS) injection in hemiplegic shoulder pain?

1.3 Significance of this study

SSNB is an effective and safe method for pain relief and increases ROM in many group of patients who had shoulder pain such as non specific shoulder pain (5),chronic shoulder pain(6) and rotator cuff tendinitis(7). SSNB can be performed using ultrasound guidance where injection of Bupivacaine is made at posterior shoulder towards suprascapular notch. Side effects include; worsening pain, soreness, bruising, nerve damage, allergic reaction.

IAS on the other hand is performed by injecting 40 mg of Triamcinolone Acetonide along with 2 ml of Lidocaine 1% into glenohumeral articular space (8). Systematic reviews of treatments for sub acromial pain favor IAS over the following options: ergonomic changes, NSAID, acupuncture, ROM and strengthening exercises, ultrasound, ice, heat, and physical therapy (9,10). Side effects include; post injection flare, disturbance of menstrual pattern, facial flushing, subcutaneous tissue atrophy, skin depigmentation, infection, and tendon rupture (13).

2 studies done so far that compare IAS vs SSNB head to head; Yasar et al,2011 and Jeon et al, 2014 only followed up the patients up to 1/12 only. Besides, there was no functional outcome measure done (11,12). Other study done with longer follow up times such as Adey-Wakeling et al, 2013 SSNB vs s/c saline (Placebo) consistently demonstrated superior, statistically significant pain reduction compared with s/c saline (placebo) even at 12/52 post injection (13).

Another randomized controlled trial (RCT) by Rah et al,2012 in comparing IAS vs subacromial lignocaine (placebo) showed significant improvement of visual analogue scale (VAS)-day/night, ROM as well as SDQ, in the treatment group even at 8/52(14). Besides, stroke is extremely common in Malaysia and is the 3rd leading cause of death in our country. Stroke patients in Malaysia is generally younger with mean age of stroke onset between 54.5 and 62.6 (15).

HSP will affect stroke recovery as the pain interfere with rehabilitation and has a potential to worsen the disability in hemiplegic patients and negatively impaired quality of life (QOL) (16).

2.0 Methodology

2.1 Study Design

This study design is prospective, double blinded interventional study. In this study, patient will be blinded from the interventions they are receiving; intraarticular steroid injection or supra-scapular nerve block. Investigator that will be assessor will also be blinded from knowing the interventions that patients received.

2.1.1 Enrollment Patients referred to SMART Clinic for hemiplegic shoulder pain will be examined and recruited. Patients who did not fulfill the inclusion and exclusion criteria will be excluded.

Numerical rating score (NRS) pain score at maximum passive ROM of shoulder flexion, abduction, internal and external rotation, Maximum passive ROM of shoulder flexion, abduction, internal and external rotation, Shoulder Pain and Disability Index (SPADI) and Shoulder Disability Questionnaire (SDQ) will be measured prior to intervention.

2.1.2 Allocation The patients recruited will then be randomly allocated using a randomization computer program into 2 separate groups; Suprascapular nerve block(SSNB) group and Intraarticular steroid(IAS) group. The assessor and patients are blinded to the type of intervention the patient is receiving. The injector who is a skilled interventionist will not be blinded.

2.1.3 Intervention Suprascapular nerve block (SSNB) and Intraaticular steoid(IAS) injection will be performed by skilled interventionist.

2.1.4 Evaluations Numerical rating score (NRS) pain score at maximum passive ROM of shoulder flexion, abduction, internal and external rotation and maximum passive ROM of shoulder flexion, abduction, internal and external rotation will be assessed and recorded at 1 hour, 1 month and 3 months after intervention. Shoulder Pain and Disability Index (SPADI) and Shoulder Disability Questionnaire (SDQ) will be measured at 1 month and 3 months post intervention.

2.2 Setting

• Rehabilitation Clinic, University of Malaya Medical Center (UMMC)

2.3 Sample Size

A power analysis program G* Power was used to calculate the sample size. The effect size of study by Jeon et al is 0.3. With the power of study set at 0.8 and alpha set at 0.05, the sample size for this study based on G* Power sample size calculator is set at 64; 32 each arm. However, to allow for 25% attrition rate, the sample size is set at 86; 43 each arm.

3.0 Data Collection Methods

Primary Outcome :

* Numerical rating score (NRS) pain score at maximum passive ROM of shoulder flexion, abduction, internal and external rotation
* To be collected at baseline, 1 hour, 1 month and 3 months post injection

Secondary outcome :

* Maximum passive ROM of shoulder flexion, abduction, internal and external rotation
* Measured at baseline, 1 hour, 1 month and 3 months post injection.
* Shoulder Pain and Disability Index (SPADI) and Shoulder Disability Questionnaire (SDQ)
* Measured at baseline, 1 month and 3 months post intervention.
* Using face to face interview

3.1 Data Analysis

Data from this study will be analysed using Statistical Package for Social Science (SPSS) software.

Demographics of 2 groups will be analyzed using Mann-Whitney U tests and Chi-Square test of association.

Primary objective:

Pain reduction:

Pre-post intervention intra-group; post-intervention inter-group: paired t-test

Secondary objectives:

ROM improvement: pre-post intragroup; post-intervention inter-group: paired t-test and analysis of variance (ANOVA)

Functional improvement of SDQ and SPADI: pre-post intra-group; post-intervention inter-group: paired t-test

4.0 Strength and Limitation

Strength

* Secondary outcomes include functional outcomes such as SPADI Score and SDQ
* Longer follow up period at 3 months compared to study by Jeon et al and Yasar et al at 1 month
* Bigger sample size Limitation
* Single center study
* Risk of patient loss to follow-up
* Recruitment will be a challenge

ELIGIBILITY:
Inclusion Criteria:

* Brain lesion recognized by CT Brain scan or MRI brain
* Hemiplegic shoulder pain of at least 2 weeks in duration
* Failed standard treatment with oral medications and physical modalities
* Age 20-70 years old
* Pain score of at least numerical rating scale (NRS) 3/10 at movement
* Mini Mental State Examination(MMSE) at least 24/30

Exclusion Criteria:

* Neuropathic pain
* Severe aphasia affecting communication
* Previous trauma history to affected shoulder and preexisting shoulder pain/pathology
* Previous shoulder injection within the past 3 months

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2019-07-11 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Numerical rating score (NRS) pain score at maximum passive range of motion (ROM) of shoulder flexion, abduction, internal and external rotation | To be collected at baseline, 1 hour, 1 month and 3 months post injection
  The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).

SECONDARY OUTCOMES:
Changes in maximum passive ROM of affected shoulder flexion, abduction, internal and external rotation | Measured at baseline, 1 hour, 1 month and 3 months post injection.
  Measured by assessor who is blinded to the intervention in supine position.
Shoulder Pain and Disability Index (SPADI) | Measured at baseline, 1 month and 3 months post intervention. *SPADI not measured at 1 hour post injection as functional outcome measure are not expected to change within 1 hour.
  Shoulder Pain and Disability Index (SPADI) was developed to assess pain and disability related to shoulder problems.
  Pain dimension has 5 questions regarding the pain severity. Disability components are assessed with 8 questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use.
  Every question is given a scale from 0 to 10.
  For Pain component, 0 = no pain and 10 = the worst pain imaginable For disability component, 0 = no difficulty and 10 = so difficult that it requires help.
  The total score from both components will be divided by 130 X 100 and will be in percentage.
  The higher the score indicates the worse outcome.
Shoulder Disability Questionnaire (SDQ) | Measured at baseline, 1 month and 3 months post intervention. *SDQ not measured at 1 hour post injection as it requires the patient to answer questions regarding the painful shoulder in the preceding 24 hours
  It contains 16 items describing common situations that may induce symptoms in patients with shoulder disorders. All items refer to the preceding 24 hours.
  It is a useful instrument to assess functional disability in longitudinal studies
  The 16 questions requires Yes or No answer. The total Yes will then be divided by 16 X 100 and will be in percentage.
  The higher the marks, the greater the disability is and indicates the worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: ANWAR BIN SUHAIMI, MBBS, Principal Investigator — SENIOR LECTURER AND REHABILITATION PHYSICIAN; SOO CHIN CHAN, MBBS, Principal Investigator — LECTURER AND REHABILITATION PHYSICIAN
Locations (1):
- Rehabilitation Medicine Clinic, Pusat Perubatan Universiti Malaya,, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langhorne P, Stott DJ, Robertson L, MacDonald J, Jones L, McAlpine C, Dick F, Taylor GS, Murray G. Medical complications after stroke: a multicenter study. Stroke. 2000 Jun;31(6):1223-9. doi: 10.1161/01.str.31.6.1223. PMID 10835436
- [Background] Poduri KR. Shoulder pain in stroke patients and its effects on rehabilitation. J Stroke Cerebrovasc Dis. 1993;3(4):261-6. doi: 10.1016/S1052-3057(10)80071-0. Epub 2010 Jun 8. PMID 26487463
- [Background] Viana R, Pereira S, Mehta S, Miller T, Teasell R. Evidence for therapeutic interventions for hemiplegic shoulder pain during the chronic stage of stroke: a review. Top Stroke Rehabil. 2012 Nov-Dec;19(6):514-22. doi: 10.1310/tsr1906-514. PMID 23192716
- [Background] Caglar NS, Akin T, Aytekin E, Komut EA, Ustabasioglu F, Okur S, Dogan Y, Erdem HI, Ataoglu E, Yalcinkaya E. Pain syndromes in hemiplegic patients and their effects on rehabilitation results. J Phys Ther Sci. 2016 Mar;28(3):731-7. doi: 10.1589/jpts.28.731. Epub 2016 Mar 31. PMID 27134349
- [Background] Taskaynatan MA, Yilmaz B, Ozgul A, Yazicioglu K, Kalyon TA. Suprascapular nerve block versus steroid injection for non-specific shoulder pain. Tohoku J Exp Med. 2005 Jan;205(1):19-25. doi: 10.1620/tjem.205.19. PMID 15635270
- [Background] Shanahan EM, Ahern M, Smith M, Wetherall M, Bresnihan B, FitzGerald O. Suprascapular nerve block (using bupivacaine and methylprednisolone acetate) in chronic shoulder pain. Ann Rheum Dis. 2003 May;62(5):400-6. doi: 10.1136/ard.62.5.400. PMID 12695149
- [Background] Di Lorenzo L, Pappagallo M, Gimigliano R, Palmieri E, Saviano E, Bello A, Forte A, DeBlasio E, Trombetti C. Pain relief in early rehabilitation of rotator cuff tendinitis: any role for indirect suprascapular nerve block? Eura Medicophys. 2006 Sep;42(3):195-204. PMID 17039215
- [Background] Buchbinder R, Green S, Youd JM. Corticosteroid injections for shoulder pain. Cochrane Database Syst Rev. 2003;2003(1):CD004016. doi: 10.1002/14651858.CD004016. PMID 12535501
- [Background] Johansson K, Oberg B, Adolfsson L, Foldevi M. A combination of systematic review and clinicians' beliefs in interventions for subacromial pain. Br J Gen Pract. 2002 Feb;52(475):145-52. PMID 11885825
- [Background] Adey-Wakeling Z, Liu E, Crotty M, Leyden J, Kleinig T, Anderson CS, Newbury J. Hemiplegic Shoulder Pain Reduces Quality of Life After Acute Stroke: A Prospective Population-Based Study. Am J Phys Med Rehabil. 2016 Oct;95(10):758-63. doi: 10.1097/PHM.0000000000000496. PMID 27003204
- [Background] Rah UW, Yoon SH, Moon DJ, Kwack KS, Hong JY, Lim YC, Joen B. Subacromial corticosteroid injection on poststroke hemiplegic shoulder pain: a randomized, triple-blind, placebo-controlled trial. Arch Phys Med Rehabil. 2012 Jun;93(6):949-56. doi: 10.1016/j.apmr.2012.02.002. Epub 2012 Apr 5. PMID 22483593
- [Background] Chae J, Mascarenhas D, Yu DT, Kirsteins A, Elovic EP, Flanagan SR, Harvey RL, Zorowitz RD, Fang ZP. Poststroke shoulder pain: its relationship to motor impairment, activity limitation, and quality of life. Arch Phys Med Rehabil. 2007 Mar;88(3):298-301. doi: 10.1016/j.apmr.2006.12.007. PMID 17321820
- [Result] Yasar E, Vural D, Safaz I, Balaban B, Yilmaz B, Goktepe AS, Alaca R. Which treatment approach is better for hemiplegic shoulder pain in stroke patients: intra-articular steroid or suprascapular nerve block? A randomized controlled trial. Clin Rehabil. 2011 Jan;25(1):60-8. doi: 10.1177/0269215510380827. Epub 2010 Oct 13. PMID 20943716
- [Result] Jeon WH, Park GW, Jeong HJ, Sim YJ. The Comparison of Effects of Suprascapular Nerve Block, Intra-articular Steroid Injection, and a Combination Therapy on Hemiplegic Shoulder Pain: Pilot Study. Ann Rehabil Med. 2014 Apr;38(2):167-73. doi: 10.5535/arm.2014.38.2.167. Epub 2014 Apr 29. PMID 24855610